CLINICAL TRIAL: NCT05253196
Title: Enema Device for Children With Spina Bifida
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-2976
Record Dates: First submitted 2021-09-13; First posted 2022-02-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Spina Bifida; Fecal Incontinence
MeSH Terms: conditions — Spinal Dysraphism; Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of Foley Catheter Assistive Device (Experimental): All participants will use Foley Catheter Assistive Device
  Interventions: Device: Use of the foley catheter assistive device

INTERVENTIONS:
Device: Use of the foley catheter assistive device — All participants will use the foley catheter assistive device when performing their daily enema

SUMMARY:
The International Center for Colorectal and Urogenital Care at Children's Hospital Colorado treats patients who suffer from many different colorectal issues such as anorectal malformation, Hirschsprung disease, and severe constipation. Many of these patients suffer from fecal incontinence. The investigators have developed a week long bowel management program (BMP) that is offered every month to help these kids stay clean of stool in the underwear, by finding the perfect enema recipe to clean the colon for 24 hours. This allows one to perform an enema once every day, clean their colon, and remain free of 'accidents'. Many spina bifida patients also suffer from fecal incontinence and are referred to this BMP. The overall success rate for all patients who suffer from fecal incontinence is 95%, however the success rate for spina bifida patients is only 77%. The reason for this decrease in success is due to the lack of anal sphincter tone in spina bifida patients, which leads to inadvertent leakage and spillage of enema fluid and bowel content during enema administration. The purpose of this study is to create and test an enema administration device that improves upon current methods.

DETAILED DESCRIPTION:
Patients meeting inclusion criteria will be enrolled while they are here on campus for a regular clinic visit. Once they consent, they will complete a baseline survey, and will be given the FCAD with the instruction manual and the investigators will go over how to use the device and answer any questions. The PI will be available throughout the study for any questions that may arise. Participants will use the device for their regular enemas for up to 4 weeks. If the device is negatively impacting enema administration, they can choose to stop using the device at any time but it is preferable that participants use the device five times before they decide it is not working for them. Once a participant has used the device for 4 weeks or has chosen to opt out of completing the 4-week trial, they will complete a second survey. The baseline survey will assess how current enema administration practices are going and the second survey will assess how well enema administration is going while using the device. If time allows and user feedback indicates a need, the device will be modified, and participants asked to use the second version for up to 4 weeks. Again, if the device is negatively impacting enema administration, they can choose to stop using the second version of the device at any time but it's preferable that participants use it five times before deciding it is not working for them. Once a participant has used the second version of the device for 4 weeks, or chosen to opt out of completing the 4-week trial, they will complete a third survey assessing the second version of the device. If traveling to CHCO is not convenient, the second version of the device will be mailed to the participant and they will complete the surveys via email or over the phone. This eliminates the need for a return trip to CHCO. REDCap will be used for all surveys. If participants are not able to complete the surveys electronically for any reason, they will complete a hardcopy version, or the survey will be administered over the phone, whichever is convenient for the participant.

ELIGIBILITY:
Inclusion Criteria:

* Poor sphincter tone
* Perform regular enemas for bowel management (due to fecal incontinence)
* 2 - 30 years old

Exclusion Criteria:

* Non English speakers
* Prisoners
* Pregnant women
* Wards of state
* Decisionally challenged adults

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Feedback Survey | 4 Weeks
  All participants will complete a feedback survey at baseline to assess satisfaction with current enema administration and again after using the device to determine if the device improves enema administration process. Each question from baseline will be compared to the same question after use of device to determine if the response is more positive with device use.

IPD SHARING:
Plan to Share IPD: No